CLINICAL TRIAL: NCT00361400
Title: Combined Hormonal Contraceptive Use in High Risk Women: A Longitudinal Study
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Other Study IDs: R01HD045480-03 (NIH)
Record Dates: First submitted 2006-08-04; First posted 2006-08-08 (Estimated); Last update posted 2013-08-02 (Estimated); Status verified 2013-08

CONDITIONS: Pregnancy
Keywords: pregnancy; hormonal contraception

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — urine for pregnancy testing

SUMMARY:
This study is an examination of "high risk" young women, 15-24 years of age, who initiate first time use of vaginal ring, oral contraceptives, contraceptive path, or Depo-provera.

DETAILED DESCRIPTION:
Approximately 1600 young women will be enrolled in a 12 month, observation study of their contraceptive use. They will complete surveys at baseline, 3, 6 and 12 months. They will also undergo pregnancy testing at baseline, 6 and 12 month visits. The study is examining such things are the relationship between partnerships, parental and peer influences, and contraceptive choice; Factors associated with long term continuation of contraceptive methods; Attributes of new hormonal contraceptive associated with user satisfaction and long-term continuation; And the extent to which high-risk women who use these methods are also condom users and determine the characteristics of these users.

ELIGIBILITY:
Inclusion Criteria:

- 15-24 years old, English or spanish speaking, Starting ring, pill, patch, or Depo for first time, Sexually active, Single, Not pregnant, Living in Bay Area for next 12 months

Exclusion Criteria:

Past user of method, Married, Pregnant, Moving out of area, Not sexually active

Ages: 15 Years to 24 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Planned Parenthood patients who present to start a hormonal birth control for the first time.
Sampling Method: Non-Probability Sample
Enrollment: 1387 (Actual)
Dates: Start 2005-08; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tina R Raine, MD, MPH, Principal Investigator — University of California, San Francisco; Cynthia Harper, PhD, Principal Investigator — University of California, San Francisco
Locations (5):
- United States (5):
  - Planned Parenthood-Golden Gate, Hayward, California
  - Planned Parenthood-Golden Gate, Oakland, California
  - Planned Parenthood - Shasta Diablo, Richmond, California
  - University of California, San Francisco, San Francisco, California
  - Planned Parenthood - Shasta Diablo, Vallejo, California

REFERENCES:
- See also: Related Info — http://www.ncbi.nlm.nih.gov/pmc/articles/PMC3154007/